CLINICAL TRIAL: NCT06722092
Title: Can Immersive Virtual Reality Magnify Treatment Outcomes of Script Training on Cantonese Speakers with Chronic Aphasia: a Randomized Controlled Trial
Brief Title: VR and Scrip Training of PWA, Randomized Controlled Trial
Acronym: VRSTPWA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Prof FONG NAI KUEN KENNETH (Unknown); Dr LI SHI PUI (Unknown); Dr NG HIU FUNG PETER (Unknown); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20230228003-01
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-08

CONDITIONS: Aphasia, Acquired; Chronic Stroke
Keywords: functional communication; randomized controlled trial; script training; immersive reality; aphasia intervention
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VR-based script training (Experimental)
  Interventions: Behavioral: VR-based script training
- Control (No Intervention)
- Computerized script training without VR (Active Comparator)
  Interventions: Behavioral: Conventional script training

INTERVENTIONS:
Behavioral: VR-based script training — The PWA will wear a head-mounted VR device (e.g., Metaverse Oculus Quest 2 or other commercially available devices) for 30 minutes, which intends to create an immersive environment for training. Scripts trained in the computerized script training program in a particular session will be practiced. Cinematic 360˚ photo-real scenarios of daily contexts such as a restaurant or a grocery store will be displayed in the device while a communication partner, e.g., a waiter in the restaurant or a shopkeeper of a grocery store will initiate the conversation by producing the corresponding part of the script. The PWA will be given time to respond. Upon the completion of PWA's respond, the next conversational turn will be initiated. The clinical assistant, who accompanies the PWA in the entire training session, will control the flow of the 360 ˚ videos.
  Arms: VR-based script training
Behavioral: Conventional script training — The flow of training is identical to the VR condition, except that photos depicting the scenarios and prerecorded conversational turns will be presented to the PWA on a computer screen with the same procedures mentioned in the VR condition.
  Arms: Computerized script training without VR

SUMMARY:
The goal of this RCT is to investigate if computerized script training may promote functional communication and nonverbal cognitive functions of Cantonese-speaking PWA, and whether VR may further magnify the treatment outcomes.

The main research questions are:

1. Can script training promote verbal functional communication of Cantonese-speaking PWA?
2. Can script training enhance nonverbal cognitive functions of Cantonese-speaking PWA?
3. Can VR magnify verbal and nonverbal treatment outcomes of script training of PWA?

ELIGIBILITY:
Inclusion Criteria:

1. a stroke onset more than six months, with an Aphasia Quotient (AQ) below 96.4, as evaluated by the Cantonese version of Western Aphasia Battery (CAB; Yiu, 1992),
2. premorbid fluent Cantonese speakers,
3. aged between 30 and 80 years,
4. no reported progressive neurogenic disorders such as dementia or Parkinson's disease,
5. no motor speech disorders of moderate to severe level, and
6. normal or corrected-to-normal vision and hearing functions

Exclusion Criteria:

1. concurrent participation in other aphasia treatment trials, and
2. incompatibility with immersive VR exposure such as complains of nausea, headache, or other severe discomforts during trial use of a head-mounted device during screening.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Percentage accuracy of treatment probe correctly produced | From baseline up to 8-week post training
  Participant's production accuracy of the trained scripts in read-aloud and no-cue conditions.
Time to produce each of the scripts in the treatment probe | From baseline up to 8-week post training
  Participant's production time of the trained scripts in read-aloud and no-cue conditions.
Number of sessions to reach performance criteria in session probe | From baseline up to 8-week post training

SECONDARY OUTCOMES:
Cantonese version of the Western Aphasia Battery (CAB) to measure aphasia severity | From baseline up to 8-week post training
Cantonese version of the Amsterdam-Nijmegen Everyday Language Test to measure verbal communication effectiveness in conversation via 20 culturally appropriate scenarios | From baseline up to 8-week post training
Cantonese version of the 20-item Communication Outcome after Stroke (Can-COAST) as a self-reported outcome on communication and quality of life | From baseline up to 8-week post training
  The questionnaire consists of 20 questions, and participants will be asked to evaluate their functional communication and quality of life based on a 5-point Likert scale. Higher scores reflect better functional communication performance and quality of life.
Subtest 1 (map search) and 3 (elevator counting) of Test of Everyday Attention to assess attention | From baseline up to 8-week post training
  The sub-test 1 aims to tap sustained and selective visual attention via identifying the target symbol in a map while the sub-test 3 assesses auditory selective attention via counting the number of target tones in the presence of distractors with different tones.
Digit span forward and backward task to assess verbal short-term and working memory | From baseline up to 8-week post training
  The longest span of participant correctly recalled in the digit span forward and backward task.
Test of Nonverbal Intelligence-third edition (TONI-3) to assess executive function | From baseline up to 8-week post training
  A norm-referenced test that uses abstract figures to evaluate abstract reasoning and problem-solving.
Wisconsin Card Sort Test (WCST) to assess executive function | From baseline up to 8-week post training
  WCST assesses cognitive flexibility and reasoning via matching cards with respect to color, quantity, and shape upon different rules and feedback given.

CONTACTS AND LOCATIONS:
Overall Officials: Winsy WS Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: Yes
The IPD, together with the study protocol, will be shared in an open-access data repository (e.g., OSF).
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared starting from three months after manuscript publication.
Access Criteria: The IPD and study protocol will be shared in an open-access data repository without restrictions.